CLINICAL TRIAL: NCT06987149
Title: Prefabricated CAD/CAM Zirconia Membrane Versus Contour Augmentation Simultaneously With Dental Implant Placement in the Anterior Esthetic Area.
Brief Title: A Randomized Controlled Trial Evaluating Dental Implant Placement in the Anterior Esthetic Zone Using Two Guided Bone Regeneration Techniques: Prefabricated CAD/CAM Zirconia Membrane vs. Contour Augmentation.
Acronym: RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammed Mashhout Eisa Anas (Other)
Responsible Party: Sponsor-Investigator, Mohammed Mashhout Eisa Anas, Dentist, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OMPDR 5-23 2
Record Dates: First submitted 2025-05-14; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2024-05

CONDITIONS: Alveolar Ridge Augmentation, Dental Implants; Alveolar Ridge Deficiency in the Anterior Esthetic Zone
Keywords: Alveolar ridge augmentation; Dental implant; Guided bone regeneration; Countour augmentation; Prefabricated CAD/CAM zirconia membrane; Alveolar ridge deficiency; Anterior Esthetic Zone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CAD/CAM Zirconia Membrane Group (Experimental): Participants in this group will undergo guided bone regeneration using a customized, prefabricated CAD/CAM zirconia membrane designed based on the individual's ridge defect morphology. This membrane will be used in combination with particulate bone graft material and placed simultaneously with the dental implant in the anterior maxilla.
  Interventions: Device: CAD/CAM Zirconia Membrane
- Contour Augmentation Group (Active Comparator): Participants in this group will undergo conventional guided bone regeneration using particulate bone graft material covered with a resorbable collagen membrane. The grafting procedure will be performed simultaneously with dental implant placement in the anterior maxilla.
  Interventions: Procedure: Contour Augmentation

INTERVENTIONS:
Device: CAD/CAM Zirconia Membrane — A prefabricated, non-resorbable zirconia membrane fabricated using CAD/CAM technology for guided bone regeneration in horizontal ridge deficiencies during simultaneous dental implant placement.
  Arms: CAD/CAM Zirconia Membrane Group
Procedure: Contour Augmentation — Traditional guided bone regeneration using particulate bone graft and a resorbable collagen membrane, placed concurrently with the dental implant to augment horizontal ridge deficiencies.
  Arms: Contour Augmentation Group

SUMMARY:
This clinical trial aims to compare two guided bone regeneration (GBR) techniques in patients with horizontal ridge deficiency in the anterior esthetic region. Specifically, it evaluates the use of a prefabricated CAD/CAM zirconia membrane versus conventional contour augmentation performed simultaneously with dental implant placement. The study includes male and female patients aged 20 to 50 years who are in good general health, maintain adequate oral hygiene, and present with a Class I ridge defect as per Seibert's classification.

The primary objective is to determine whether the customized zirconia membrane provides equivalent clinical and radiographic outcomes in terms of bone gain and soft tissue healing compared to the contour augmentation technique. Participants will also report their postoperative discomfort and overall satisfaction using a 100-point visual analog scale (VAS), recorded at multiple time points: 1, 6, and 12 hours, as well as 1, 3, 7, and 15 days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders within the age range of 20-50 years.
* Patients with good general health and adequate oral hygiene practices.
* Stable periodontal condition and favorable soft tissue profile.
* Alveolar ridge that has a Class I defect according to Seibert's classification of ridge defects.

Exclusion Criteria:

* Patients with medical conditions or systemic diseases precluding periodontal surgery or hampering wound healing (e.g., uncontrolled diabetes mellitus or metabolic bone disorders).
* Patients subjected to irradiation in the head and neck area.
* Patients with a history of taking any medications in the previous 6 months that may interfere with periodontal tissue health or healing.
* Patients have poor oral hygiene and motivation.
* Patients with active periodontitis or acute infection in the area intended for implant placement.
* Females who are pregnant or trying to conceive, and nursing mothers.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Alveolar bone gain in millimetres (mm) in the edentulous alveolar ridge | Six months
  Assessment of the horizontal and vertical bone gain in millimetres (mm) in the edentulous alveolar ridge from baseline (implant placement and grafting) to six months after surgery.

SECONDARY OUTCOMES:
Periodontal Soft Tissue Healing (Modified Wound Healing Index - MWHI) | Baseline (day of surgery), and postoperatively at 4, 8, 12, and 24 weeks
  Evaluation of periodontal soft tissue healing around the surgical site using the Modified Wound Healing Index (MWHI) developed by Huang et al. This index categorizes wound healing based on clinical parameters including mucosal edema, erythema, graft exposure, and presence of suppuration. Scores range from 1 to 3:
  Score 1 - Uneventful Healing: No or minimal mucosal edema or erythema, with no suppuration or graft exposure.
  Score 2 - Normal Healing: Slight to moderate mucosal edema, erythema, and/or graft exposure, but without suppuration.
  Score 3 - Poor Healing: Significant mucosal edema, erythema, graft exposure, and presence of suppuration.
Patient-Reported Postoperative Discomfort and Satisfaction | 1 hour, 6 hours, 12 hours, and 1, 3, 7, 15 days postoperatively
  Assessment of postoperative discomfort and overall patient satisfaction using a 100-point Visual Analog Scale (VAS). Participants will self-report their pain levels and satisfaction at multiple postoperative time points: 1, 6, and 12 hours, as well as 1, 3, 7, and 15 days after surgery.
Membrane-Related Operative Time | Recorded during the implant placement and bone regeneration surgery
  Measurement of the time (in minutes) required to place the guided bone regeneration membrane during the surgical procedure. This will assess the efficiency and ease of use of the prefabricated CAD/CAM zirconia membrane compared to conventional contour augmentation.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry- Tanta university, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided